CLINICAL TRIAL: NCT02796222
Title: Factor Product Utilization and Health Outcomes in Patients With Hemophilia A and B in Canada: An Observational Study of Real-world Outcomes
Brief Title: Factor Product Utilization and Health Outcomes in Patients With Hemophilia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Shannon Jackson, Clinical Associate Professor, University of British Columbia
Other Study IDs: CAN-FAB-15-10911
Record Dates: First submitted 2016-05-26; First posted 2016-06-10 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A, Congenital; Hemophilia B, Congenital
Keywords: Hemophilia; Recombinant factor VIII; Recombinant factor VIII Fc; Recombinant factor IX; Patient-reported outcomes; Recombinant factor IX Fc
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hemophilia A patients on rFVIIIFc: Patients with hemophilia A who switch from on-demand or prophylactic treatment with rFVIII to rFVIIIFc
- Hemophilia A patients on rFVIII: Patients with hemophilia A who remain on on-demand or prophylactic treatment with rFVIII
- Hemophilia B patients on rFIXFc: Patients with hemophilia B who switch from on-demand or prophylactic treatment with rFIX to rFIXFc
- Hemophilia A patients on rFIX: Patients with hemophilia B who remain on on-demand or prophylactic treatment with rFIX

SUMMARY:
Recombinant factor VIII Fc (rFVIIIFc) and recombinant factor IX Fc (rFIXFc) are extended half-life coagulation factors approved by Health Canada in 2014 for the treatment of severe hemophilia A and B, respectively. The objectives of this observational study is to describe the change in annual factor consumption, clinical and patient-reported outcomes for patients who switch from recombinant factor VIII (rFVIII) and recombinant factor IX (rFIX) to rFVIIIFc/ rFIXFc in Canada, and to explore clinicians' and patients' reasons for switching or not switching.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥12 years of age with severe and moderate congenital hemophilia A or B (baseline factor activity<5%)
2. Ability to understand the purpose and risks of the study and provide signed and dated informed consent or assent and authorization to use protected health information (PHI) in accordance with national and local privacy regulations.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Patients with an existing bleeding disorder other than hemophilia A or B
3. History of hypersensitivity or severe allergic reactions to factor products
4. Patients currently participating in a phase 1-3 study with another factor replacement product
5. Unable to adhere to the study requirements based on the judgment of the Prescribing Physician (e.g. unable to enter accurate and timely infusion and bleeding records)

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted in male patients ≥12 years of age with severe and moderate hemophilia A or hemophilia B (baseline factor level <5%) who are able to sign the informed consent or assent.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Change in the total annualized factor consumption (in units/kilogram/year) | From baseline to 24-month period on rFVIIIFc or rFIXFc

SECONDARY OUTCOMES:
Change in health-related quality of life (HRQoL) SF-36 | From baseline to 3 months, 12 months and 24 months
  HRQoL will be measured using Short Form 36 (SF-36) in all patients
Change in health-related quality of life (HRQoL) Haem-A-Qol | From baseline to 3 months, 12 months and 24 months
  Haem-A-QoL in patients over age 18 years
Change in health-related quality of life (HRQoL) CHO-KLAT | From baseline to 3 months, 12 months and 24 months
  The Canadian Hemophilia Outcomes- Kids Life Assessment Tool (CHO-KLAT) in patients between ages 13-18 years
Change in the Work Productivity and Impairment Questionnaire (WPAI+CIQ: HS) score | From baseline to 3 months, 12 months and 24 months
Change in chronic pain Numeric Rating Scale (0-10) | From baseline to 3 months, 12 months and 24 months
Change in chronic pain "Bodily Pain" subscale of SF-36 | From baseline to 3 months, 12 months and 24 months
Change in physical activity (IPAQ) | From baseline to 3 months, 12 months and 24 months
  Physical activity will be measured using the International Physical Activity Questionnaire (IPAQ)
Change in physical activity "Physical Functioning" subscale of SF-36. | From baseline to 3 months, 12 months and 24 months
Change in treatment satisfaction "Treatment" domain of Haem-A-QoL | From baseline to 3 months, 12 months and 24 months
Change in treatment satisfaction abbreviated 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) questionnaire. | From baseline to 3 months, 12 months and 24 months
  Abbreviated 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) questionnaire.
Change in mood "Mental Health" subscale of SF-36 | From baseline to 3 months, 12 months and 24 months
  partner or caregiver's subjective assessment of subject's mood from baseline to 3 months.
Change in mood partner/caregiver subjective assessment numeric rating scale (0-10) | From baseline to 3 months only
  Partner or caregiver's subjective assessment of subject's mood from baseline to 3 months.
Clinicians' and patients' reason for switching to rFVIIIFc | Baseline through study completion, an average of 2 years
  Choice among list of common reasons for changing product
Clinicians' and patients' reason for switching to rFIXFc | Baseline through study completion, an average of 2 years
  Choice among list of common reasons for changing product
Product used for treatment of breakthrough bleeding and surgical procedures | Baseline through study completion, an average of 2 years
  Choice among list of products
Total annualized number of factor infusions | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)
Annualized bleeding rate | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)
Ratio of annual factor consumption-to-annual factor prescription | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)
Number of infusions required to treat a breakthrough bleed | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)
Incremental factor utilization per joint bleed avoided | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)
  Difference in annualized factor utilization between Fc and regular non-Fc prophylaxis, divided by the difference in annualized joint bleeding rate between the two groups.
Adverse events leading to permanent discontinuation of rFVIIIFc or rFIXFc | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)
Serious adverse events | From baseline to 24-month period after product switch (or 24-month period on study for non-switchers)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Jackson, MD, Principal Investigator — Division of Hematology, Department of Medicine, University of British Columbia; Robert Klaassen, MD, Study Chair — Division of Hematology/Oncology, Department of Pediatrics, University of Ottawa; Man-Chiu Poon, MD, Study Chair — Division of Hematology, Department of Medicine, University of Calgary; Sue Robinson, MD, Study Chair — Division of Hematology, Department of Medicine, Dalhousie University; John Wu, MD, Study Chair — BC Children's hospital, Division of Hematology, Department of Medicine, University of British Columbia; Alfonso Iorio, MD, Study Chair — Hemophilia Program, Hamilton Health Services Program, McMaster University; Michelle Sholzberg, MD, Study Chair — Hemophilia Program, St. Michael's Hospital, University of Toronto
Locations (1):
- BC Hemophilia Adult Program, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No